CLINICAL TRIAL: NCT07192796
Title: Comparative Effects of Pilates and Neuromuscular Exercises on Postural Control in Dynamic Knee Valgus
Brief Title: Effects of Pilates and Neuromuscular Exercises on Postural Control in Dynamic Knee Valgus
Acronym: DKV-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şebnem Nur Alkan (Other)
Responsible Party: Sponsor-Investigator, Şebnem Nur Alkan, Assistant Professor of Physiotherapy, Atlas University, Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-22686390-050.99-41964
Record Dates: First submitted 2025-09-03; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dynamic Knee Valgus; Knee Injuries; Postural Control Deficit
Keywords: Dynamic knee valgus; Neuromuscular exercise; Pilates; Frontal plane projection angle; Postural control
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: Participants were randomized into three parallel groups: a Pilates exercise group, a neuromuscular exercise group, and a control group. Interventions were delivered over 6 weeks (18 sessions).
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind design: Both participants and the outcome assessor were blinded to group allocation. Exercise providers were not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates Exercise Group (Experimental): Participants in this group completed a 6-week supervised Pilates exercise program, with 18 sessions. The program included mat-based and resistance band exercises focusing on core stabilization and postural alignment.
  Interventions: Behavioral: Pilates Exercise Program
- Neuromuscular Exercise Group (Experimental): Participants in this group performed a progressive neuromuscular training program for 6 weeks, with 18 supervised sessions. The program emphasized balance, proprioception, dynamic stability, and strengthening of lower extremity muscles.
  Interventions: Behavioral: Neuromuscular Exercise Program
- Control Group (No Intervention): Participants in this group did not receive any exercise intervention during the 6-week period. They underwent the same baseline and post-intervention assessments as the experimental groups but continued with their usual daily activities.

INTERVENTIONS:
Behavioral: Pilates Exercise Program — A 6-week supervised Pilates exercise program, with 18 sessions. Exercises focused on core stabilization, posture, and lower limb alignment using mat-based and resistance band movements.
  Arms: Pilates Exercise Group
Behavioral: Neuromuscular Exercise Program — A 6-week supervised neuromuscular training program, 18 sessions . Training emphasized balance, proprioception, dynamic stability, and strengthening of lower extremity muscles.
  Arms: Neuromuscular Exercise Group

SUMMARY:
This randomized controlled trial aims to investigate the effects of neuromuscular and Pilates exercise programs compared with a control group in young adults with dynamic knee valgus (DKV). Thirty-six participants were randomly assigned to neuromuscular, Pilates, or control groups. The intervention groups completed a supervised exercise program three times per week for six weeks (18 sessions).

The primary outcome is the frontal plane projection angle (FPPA) during single-leg tasks. Secondary outcomes include muscle strength, balance, and vertical jump performance.

DETAILED DESCRIPTION:
This prospective, single-blind randomized controlled trial was designed to evaluate the comparative effects of Pilates and neuromuscular exercise training on lower extremity alignment and postural control in young adults with dynamic knee valgus (DKV). Ethical approval was obtained from the Istanbul Atlas University Non-Interventional Scientific Research Ethics Committee (Approval No: E-22686390-050.99-41964, 03/05/2024).

A total of 45 participants aged 18-24 years, all right-leg dominant, were initially enrolled and randomized into three groups: Pilates, neuromuscular exercise, and control (15 in each group). Randomization was performed using computerized allocation. Due to dropouts, 36 participants (12 per group) completed the study between June and August 2024.

The interventions consisted of a 6-week supervised program (18 sessions, 3 times per week). Both Pilates and neuromuscular protocols were progressive in intensity, incorporating resistance bands, core stabilization, and functional balance exercises. The control group did not receive any intervention but underwent the same baseline and post-intervention assessments.

The primary outcome was the frontal plane projection angle (FPPA) during single-leg squat and single-leg drop jump tasks, measured using 2D video analysis.

The secondary outcomes included:

Isometric strength of the gluteus medius and rectus femoris measured with a handheld dynamometer,

Balance performance assessed separately by the Biodex Postural Stability Test (overall, anterior-posterior, and medial-lateral stability indices) and the Limits of Stability Test,

Functional performance assessed by the OptoJump system, including vertical jump height, vertical jump power, and reactive strength index.

All assessments were conducted at baseline and after 6 weeks by the same physiotherapist to ensure intra-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* having asymptomatic dynamic knee valgus
* being between 18 and 24 years of age
* having no medical history, a body mass index (BMI) between 18 and 24
* no history of orthopedic, neurological, vascular, systemic, or rheumatic diseases
* no complaints of pain in any part of the body during physical activities
* the ability to communicate in Turkish (both written and verbal)

Exclusion Criteria:

* individuals with hip anteversion or retroversion or other postural disorders affecting knee kinematics, those unable to perform the exercises as demonstrated, those experiencing pain during exercises (VAS >5)
* individuals with a history of orthopedic surgery, those with strength deficits between extremities
* the presence of cognitive or psychological disorders that could hinder cooperation
* pregnancy or suspected pregnancy
* sleep disorders, regular medication use, intake of painkillers, sedatives, or psychiatric drugs within the last 24 hours
* history of chronic systemic, rheumatologic, neurological, or vascular diseases

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Frontal Plane Projection Angle (FPPA) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Participants performed a single-leg vertical drop jump from a 20 cm platform with the dominant leg while keeping their hands on the waist. Knee valgus angle at landing was recorded using 2D video analysis with a camera placed 3 m in front at a height of 45 cm.

SECONDARY OUTCOMES:
Isometric Strength of Gluteus Medius | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Isometric strength of the gluteus medius muscle was measured using the PowerTrack-II handheld dynamometer in a standardized side-lying position.
Isometric Strength of Rectus Femoris | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Isometric strength of the rectus femoris muscle was measured using the PowerTrack-II handheld dynamometer in a standardized seated position with 90° knee flexion.

OTHER OUTCOMES:
Postural Stability Test - Overall Stability Index (Biodex) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Overall stability index from the Biodex Postural Stability Test was recorded to evaluate total postural control.
Postural Stability Test - Anterior-Posterior Stability Index (Biodex) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  The anterior-posterior stability index was measured with the Biodex Postural Stability Test to assess directional balance control.
Postural Stability Test - Medial-Lateral Stability Index (Biodex) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  The medial-lateral stability index was measured with the Biodex Postural Stability Test to assess directional balance control.
Limits of Stability Test (Biodex) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Limits of Stability test measured weight-shifting ability toward illuminated targets using the Biodex Balance System.
Vertical Jump Height (OptoJump) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Vertical jump height was assessed using the OptoJump system during single-leg vertical jump tasks.
Vertical Jump Power (OptoJump) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  Vertical jump power was measured using the OptoJump system to evaluate lower extremity explosive strength.
Reactive Strength Index (RSI, OptoJump) | At baseline (Day 1) and following completion of 6 weeks of intervention (Week 6)
  RSI was calculated using the OptoJump system to assess neuromuscular efficiency during jump tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No